CLINICAL TRIAL: NCT05664243
Title: A Phase 1b / 2 Open-label Study to Investigate the Safety, Tolerance and Efficacy of Drug Resistant Immunotherapy (DRI) With Activated, Gene Modified Allogeneic or Autologous γδ T Cells (DeltEx) in Combination With Maintenance Temozolomide (TMZ) in Subjects With Recurrent or Newly Diagnosed Glioblastoma
Brief Title: A Phase 1b / 2 Drug Resistant Immunotherapy With Activated, Gene Modified Allogeneic or Autologous γδ T Cells (DeltEx) in Combination With Maintenance Temozolomide in Subjects With Recurrent or Newly Diagnosed Glioblastoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: In8bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INB-400
Record Dates: First submitted 2022-12-09; First posted 2022-12-23 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2024-10

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; Brain Neoplasms; Glioma; Neoplasms; Neuroepithelial; Central Nervous System Neoplasms; Neoplasms by Site
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms; Glioma; Neoplasms; Central Nervous System Neoplasms; Neoplasms by Site

STUDY DESIGN:
Intervention Model Description: Arm A subjects with newly diagnosed disease will receive autologously derived, genetically modified gamma-delta T cells administered with maintenance temozolomide.
  Phase 1b and Arm B subjects with relapsed disease will have allogeneic derived, genetically modified gamma-delta T cells administered with temozolomide
  Arm C subjects with newly diagnosed disease will receive allogeneic derived, genetically modified gamma-delta T cells administered with maintenance temozolomide.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- 1) Autologous Newly Diagnosed Disease: Phase 2 Arm A (Experimental): Arm A subjects with newly diagnosed disease will receive autologously derived, genetically modified gamma-delta T cells administered with maintenance temozolomide.
- 2) Allogeneic Relapsed Disease: Phase 1b and Phase 2 (Experimental): Phase 1b subjects with relapsed disease will have allogeneic derived, genetically modified gamma-delta T cells administered with temozolomide
  Interventions: Biological: Allogeneic genetically modified gamma-delta T cells
- 3) Allogeneic Newly Diagnosed Disease: Phase 2 Arm C (Experimental): Arm C subjects with newly diagnosed disease will receive allogeneic derived, genetically modified gamma-delta T cells administered with maintenance temozolomide.

INTERVENTIONS:
Biological: Autologous genetically modified gamma-delta T cells — Arm A: Cells will be administered on Day 1 of each of 6, 28-day cycles in combination with TMZ maintenance
Biological: Allogeneic genetically modified gamma-delta T cells — Phase 1b and Arm B: Cells will be administered on Day 1 of each of 6, 28-day cycles in combination with D1 of TMZ 150mg/m2
  Arms C: Cells will be administered on Day 1 of each of 6, 28-day cycles in combination with TMZ maintenance
  Arms: 2) Allogeneic Relapsed Disease: Phase 1b and Phase 2

SUMMARY:
This multicenter, Phase 1b/2 study is being conducted to determine if the experimental cell therapy is safe, tolerable and can delay the return of cancer in patients with a newly diagnosed or recurrent glioblastoma multiforme (GBM) in combination with standard chemotherapy treatment temozolomide (TMZ). If there is a 25% or greater improvement in survival in this study then the therapy should be studied further.

DETAILED DESCRIPTION:
This is a Phase 1b and 2 open-label cellular therapy trial using genetically modified gamma-delta (γδ) T cells or DeltEx Drug Resistant Immunotherapy (DRI). Gamma-delta T cells are a type of immune cell that may help the immune system recognize and kill cancer cells. The cells have been modified to make them resistant to the killing effects of chemotherapy such that they may be administered in combination with chemotherapy without being destroyed. The chemotherapy that is being used in this study is called temozolomide (TMZ) which is the standard-of-care used to treat glioblastoma patients. The DRI cells are given in combination with a standard dose of TMZ and are administered through a catheter directly into the brain where the tumor is located.

There are four arms to this study for eligible subjects with either newly diagnosed or relapsed IDH wild-type (IDH-wt) glioblastoma (GBM). Arm A will enroll newly diagnosed glioblastoma subjects to receive DRI cells derived from their own cells (autologous). The Phase 1b, Arms B and C will enroll subjects to receive DRI cells derived from a donor's cells (allogeneic). Subjects in the Phase 1b portion and Arm B must have relapsed disease, that is disease that has returned after initial treatment, while Arm A and C subjects must have newly diagnosed disease.

Prescreening subjects will have a standard-of-care surgical resection of their tumor. Once their preliminary eligibility is confirmed, they will have a Rickham catheter placed which is a device typically used to deliver chemotherapy into the brain that will be used to deliver the DRI cells directly to the tumor.

Following the surgical resection, subjects in Arm A will return to the study doctor's office/clinic to undergo a procedure called an apheresis. This procedure will isolate the immune cells from the blood to help make the DRI product for the subject. These cells include the gamma-delta T cells that will be used to make the DRI cells. Once the cells for the DRI product are made, they are frozen and stored for future use. In the Phase Ib and Arms B and C of the trial, a donor will undergo apheresis to provide the source of cells for the DRI product.

Following apheresis and confirmation that the required number of gamma-delta T cells were successfully collected; subjects in Arm A and C will begin the recommended or standard-of-care treatment for newly diagnosed GBM. This will include six weeks of chemotherapy with TMZ and radiation. Subjects will then have about a four week break prior to beginning the maintenance phase of treatment. Maintenance therapy includes five days of chemotherapy, every 28 days, which is repeated for six cycles. The previously frozen DRI product is thawed, prepared and is infused on the first day of each five-day cycle through the Rickham catheter. Subjects received a total of 6 infusions.

Subjects in the Phase Ib and Arm B will only receive one dose of TMZ along with the DRI product every 28 days for a total of six cycles.

Subjects will be observed for a of minimum 30 days after receiving the first dose of the DRI gamma-delta T cells. Subjects will be followed for potential side effects. The approximate duration of the study may be up to 15 years, or until disease progression or subjects withdraw from the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histologically or cytologically confirmed history of IDH-wild type glioblastoma

  * Phase 1b and Arm B of Phase 2: Subjects must have completed no more than one standard therapy for glioblastoma, have received no prior Avastin® therapy (unless solely used for edema management) and be eligible for resection
  * Arms A and C: Subjects must have newly diagnosed, treatment naïve glioblastoma
  * Phase 1b and Arm B and Arm C: Subjects must have a partially matched haploidentical or matched related donor.
* Subjects with magnetic resonance imaging (MRI) features consistent with and suspicious for recurrent malignant glioma in Phase 1b and Arm B.
* Agreeable to inserting and maintaining a Rickham catheter.
* ≥ 18 years of age.
* Karnofsky Performance Status ≥ 70%
* Female subjects of childbearing potential must have a negative urine/serum pregnancy test within 72 hours of study enrollment. Female subjects of childbearing potential are those who have not been surgically sterilized or have not been free of menses for > 2 years.
* Male subjects and their female partners and female subjects of childbearing potential must be willing to use a combination of two methods of birth control or be surgically sterile or abstain from heterosexual activity for the course of the study.

Exclusion Criteria:

* Subject in Arm A or donor from Phase 1b, Arms B, and Arm C received vaccinations within 4 weeks or underwent surgery (major or minor) within 72 hours before leukapheresis collection.
* Cellular immunotherapy or gene therapy or within six weeks prior to entering the study, surgical resection or alkylating agent chemotherapy within four weeks prior to entering the study, receiving tumor treating fields (TTF) Optune therapy, or have received experimental immunotherapy at any time
* Subjects receiving any other investigational agents concurrently while on study.
* Have not recovered from adverse events (≤ Grade 1) from previously administered therapy. Subjects with alopecia unless of immune origin are an exception to this criterion and may qualify for this study
* Have received prior treatment with an allogeneic therapy, including bone marrow or solid tumor transplant.
* Concurrent malignancy or an active second malignancy. Subjects with a history of second malignancy must have no evidence of cancer for two years prior to enrolment or have a surgically cured cancer with low risk of recurrence to enroll. Discuss with medical monitor prior to enrolment.
* Contraindication to the placement of an intracranial access device (Rickham catheter) at the time of surgery.
* Prior history of encephalitis, multiple sclerosis, or other CNS infection <1 year prior to glioblastoma diagnosis.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, or any other medical condition that precludes surgery. Also, medical/surgical/psychiatric illness/social situations that would limit compliance with study requirements or confound interpretation of safety and efficacy data. Subjects with a history of seizure as a result of their glioblastoma must be seizure free and on appropriate anti-epileptic medication for 3 weeks prior to dosing with the investigational agent.
* Allergies/hypersensitivity to amino bisphosphonates such as Zoledronate®, Pamidronate® or similar.
* History of HIV or active hepatitis even if well controlled or history of an autoimmune condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2023-09-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Autologous Phase 2, Arm A in newly diagnosed glioblastoma: 12-month overall survival (OS) rate | 12 Months
  Date of first dose to date of death by any cause
Allogeneic Phase 1b, establishes the recommended phase 2 dose (RP2D) for phase 2 allogeneic arms and subject or product characteristics that will optimize manufacturing | 28 days
  <30% dose limiting toxicity (DLT) observed with dose
Allogeneic Phase 2, Arm B confirmed recurrent glioblastoma, 9-month overall survival (OS) | 9 Months
  Date of first dose to date of death by any cause
Allogeneic Phase 2, Arm C newly diagnosed glioblastoma, 12-month overall survival (OS) rate | 12 Months
  Date of first dose to date of death by any cause

SECONDARY OUTCOMES:
Assessment of safety | 12 Months
  Assessment of safety is based on total number of treatment emergent adverse events and serious adverse events Assessment of safety is also based on change from baseline of clinical laboratory tests including change in liver function tests, renal function and complete blood counts Assessment of safety is also based on change from baseline of vital signs including heart rate, blood pressure, temperature and pulse oximetry
Assessment of tolerability | 12 Months
  Assessment of tolerability is based on total number of treatment emergent adverse events and serious adverse events Assessment of tolerability is also based on change from baseline of clinical laboratory tests including change in liver function tests, renal function and complete blood counts Assessment of tolerability is also based on change from baseline of vital signs including heart rate, blood pressure, temperature and pulse oximetry
Overall response rate (ORR) | 12 Months
  ORR is defined as the rate of the best overall response as complete response (CR) or partial response (PR).
Time to progression (TTP) | 12 Months
  Time to progression will be defined as the time from first dose until objective tumor progression
Progression free survival (PFS) | 12 Months
  PFS will be defined as the time from first dose until objective tumor progression or death, whichever comes first.
Definition of product characteristics | 12 Months
  Product characteristics that predict for maximal success of product creation:
  Age of donor ( <50 years of age, 51-65 years of age, >65 years of age), Total white blood cell count and individual immune cell count (neutrophils, T cells, gamma delta T cells) of the apheresis product, Time to infusion of manufactured product of apheresis material (1 month, 2months)

CONTACTS AND LOCATIONS:
Overall Officials: Louis B Nabors, MD, Principal Investigator — University of Alabama at Birmingham
Locations (5):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Moffitt Cancer Center, Tampa, Florida
  - University of Louisville Hospital/James Graham Brown Cancer Center, Louisville, Kentucky
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Wexner Medical Center- James Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhao Y, Dong P, He W, Zhang J, Chen H. gammadelta T cells: Major advances in basic and clinical research in tumor immunotherapy. Chin Med J (Engl). 2024 Jan 5;137(1):21-33. doi: 10.1097/CM9.0000000000002781. Epub 2023 Aug 18. PMID 37592858